CLINICAL TRIAL: NCT00573612
Title: Exercise-based Motivational Interviewing for Fibromyalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Dr. Dennis Ang, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IRB 0708-62; R01AR054324 (NIH)
Record Dates: First submitted 2007-12-12; First posted 2007-12-14 (Estimated); Last update posted 2012-04-06 (Estimated); Status verified 2011-03

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia; Fibromyalgia patients
MeSH Terms: conditions — Fibromyalgia | interventions — Motivational Interviewing

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Placebo Comparator): Telephone Call for the Attention Control Group Each AC call will follow the same format as the MI call. During the AC call, study subjects will receive health information on important topics relevant to their illness. Specifically, there will be one topic during each phone call that includes the following: (a) overview of FMS, (b) pain, (c) fatigue (d) sleep, (e) stress, and (f) living well with FMS. The AC calls will be an avenue to transfer relevant health information from the RA to the study subject. The scheduled topics during each contact will give the call face validity (i.e., establish a credible pretense for the contact) while being neutral with respect to encouragement of exercise.
  Interventions: Behavioral: Attention Control Counseling
- 2 (Active Comparator): Telephone-delivered Motivational Interviewing Participants will receive 6 telephone calls throughout the study. Harland et al reported that the most effective intervention for promoting exercise in the primary care setting was the most intensive treatment arm that included six MI sessions (208). Importantly, in our pilot study, participants who completed 5 to 6 phone calls achieved greater symptomatic benefits than participants who had ≤ 4 phone calls. The phone calls will be scheduled at week 3, 4, 6, 8, 10 and 12 of the study. Telephone sessions may run for 30 minutes on the average
  Interventions: Behavioral: Motivational Interviewing

INTERVENTIONS:
Behavioral: Attention Control Counseling — Subjects will receive educational-based telephone counseling regarding fibromyalgia.
  Arms: 1
Behavioral: Motivational Interviewing — Subjects will receive Motivational Interviewing telephone counseling.
  Arms: 2

SUMMARY:
Fibromyalgia (FMS), defined as the presence of both chronic widespread pain and the finding of 11/18 tender points on examination, affects 2% of the general population. Drug therapy for FMS is largely symptomatic as there is not yet a complete understanding of the pathogenesis of the disease. In the past 17 years, supervised aerobic exercise has emerged as an important treatment modality to improve pain, aerobic capacity, function, and well-being. Individuals who are able to adhere to exercise almost always maintain the symptomatic benefits of exercise. Unfortunately, the rate of exercise adherence six months after the completion of a well-structured supervised exercise program is disappointingly low. Furthermore, although the efficacy of supervised aerobic exercise in the research setting is well documented, the applicability of such intervention in the clinic setting is doubtful. Therefore, we propose to conduct the Research to Encourage Exercise for Fibromyalgia (REEF), a randomized attention-controlled trial whose primary aim is to evaluate the efficacy of telephone-delivered motivational interviewing (MI) to encourage exercise, in improving exercise adherence and self-report physical function (co-primary outcome measures) for FMS patients. REEF will enroll 200 FMS patients, randomizing them to either the MI group or the attention-control (AC) group. Participants from each group will receive a total of 6 telephone calls within a 12-week period. Prior to the phone calls, participants from both groups will receive an individualized exercise prescription and 2 supervised exercise training sessions to get them started on an exercise program. All subjects will undergo comprehensive outcome assessment at baseline, week 12, week 24, and week 36. The secondary aim of this proposal is to determine the mediators between MI and improvement in self-report physical function. The proposed research is significant because our focus is the promotion of adherence to an exercise program, of adequate intensity, in order to maximize functioning and well-being for patients with FMS. The use of a predominantly home-based exercise program and telephone-delivered MI by a trained licensed practice nurse (LPN) could potentially make the proposed intervention more accessible to the greater majority of FMS patients. Furthermore, if proven efficacious, MI could readily be applied to other chronically painful conditions (e.g. chronic back pain).

ELIGIBILITY:
Inclusion Criteria:

1. American College of Rheumatology (ACR) classification criteria for FMS(203)
2. Has been on stable doses of FMS medications (i.e., cyclobenzaprine, tramadol, gabapentin, pregabalin, venlafaxine, duloxetine, pramipexole, tricyclic anti-depressant, selective serotonin reuptake inhibitor) for at least 4 weeks and willing to limit the introduction of new medications for FMS symptoms
3. Age between 18-65 years old. Because the prevalence of sub-clinical coronary artery disease increases with older age, we are excluding those who are ≥ 66 years old

Exclusion Criteria:

1. FIQ-PI score < 2
2. BPI-PS <4
3. Known cardiovascular disease, including congestive heart failure; previous episodes of angina pectoris; previous myocardial infarction; or previous revascularization procedure
4. Moderate-severe chronic obstructive pulmonary disease, including asthma
5. Uncontrolled hypertension
6. Orthopedic or musculoskeletal conditions that would prohibit moderate-intensity exercise
7. Active suicidal ideation
8. Planned elective surgery during the study period
9. Ongoing unresolved disability claims
10. Other major rheumatic conditions (i.e. rheumatoid arthritis, systemic lupus erythematosus, scleroderma and other connective tissue disease)
11. Use of medications that may affect chronotropic response to exercise, i.e. beta-blocker or calcium channel blocker
12. Pregnancy
13. Schizophrenia or other psychosis
14. Exercising 3 days a week or more. The US Surgeon General considers a physically active person as somebody who does at least 3 times a week of moderate to vigorous level of exercise(204). Thus, we are excluding the already physically active individuals from the study. In the pilot study, only 4% (2 out of 50) of the potential participants were excluded due to being physically active.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2007-12; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Measure the effects of exercise-based MI intervention improving exercise adherence. | This is a five year study, each subject will participate in a 9-month study sequence

SECONDARY OUTCOMES:
To evaluate the effects of exercise-based MI intervention in pain severity and to determine between exercise-based MI intervention and the adherence. | This is a five year study, each subject will participate in a 9-month study sequence

CONTACTS AND LOCATIONS:
Overall Officials: Dennis C. Ang, MD, Principal Investigator — Indiana University
Locations (1):
- National Institute of Fitness of Sports, IUPUI Campus, Indianapolis, Indiana, United States

REFERENCES:
- [Derived] Kaleth AS, Bigatti SM, Slaven JE, Kelly N, Ang DC. Predictors of Physical Activity in Patients With Fibromyalgia: A Path Analysis. J Clin Rheumatol. 2022 Jan 1;28(1):e203-e209. doi: 10.1097/RHU.0000000000001684. PMID 33337808
- [Derived] Kaleth AS, Slaven JE, Ang DC. Does increasing steps per day predict improvement in physical function and pain interference in adults with fibromyalgia? Arthritis Care Res (Hoboken). 2014 Dec;66(12):1887-94. doi: 10.1002/acr.22398. PMID 25049001
- [Derived] Kaleth AS, Saha CK, Jensen MP, Slaven JE, Ang DC. Effect of moderate to vigorous physical activity on long-term clinical outcomes and pain severity in fibromyalgia. Arthritis Care Res (Hoboken). 2013 Aug;65(8):1211-8. doi: 10.1002/acr.21980. PMID 23401486
- [Derived] Ang DC, Kaleth AS, Bigatti S, Mazzuca SA, Jensen MP, Hilligoss J, Slaven J, Saha C. Research to encourage exercise for fibromyalgia (REEF): use of motivational interviewing, outcomes from a randomized-controlled trial. Clin J Pain. 2013 Apr;29(4):296-304. doi: 10.1097/AJP.0b013e318254ac76. PMID 23042474